CLINICAL TRIAL: NCT02150837
Title: A Retrospective Chart Review to Assess Weight Loss in Overweight and Obese Adults Using Either the 5 & 2 & 2 Meal Replacement Plan or the 4 & 2 & 1 Meal Replacement Plan at Medifast Weight Control Centers
Brief Title: Retrospective Chart Review of the 5 & 2 & 2 and 4 & 2 & 1 Plans
Status: Completed | Type: Observational
Sponsor: Medifast, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MED 017
Record Dates: First submitted 2014-05-21; First posted 2014-05-30 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Obesity
Keywords: Obesity; Weight Loss; Meal replacements; Weight maintenance
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 5 & 2 & 2 Plan: MWCC members who used the Medifast 5 & 2 & 2 Meal Replacement Plan for weight loss.
  Interventions: Other: 5 & 2 & 2 Plan
- 4 & 2 & 1 Plan: MWCC members who used the Medifast 4 & 2 & 1 Meal Replacement Plan for weight loss.
  Interventions: Other: 4 & 2 & 1 Plan

INTERVENTIONS:
Other: 5 & 2 & 2 Plan — Medifast has developed the 5 & 2 & 2 Plan as a higher calorie and higher carbohydrate alternative. This plan may be selected for very obese (BMI ≥ 40kg/m2) or older (>65 years) individuals, or for medical (e.g., diabetes) or behavioral reasons (individuals engages in high levels of physical activity). The 5 & 2 & 2 Plan consists of 5 Medifast meal replacements, 2 Lean & Green meals, and 2 healthy snacks and provides 1,200-1,400 kcal, >72g protein, >100g of carbohydrate, and <30% of calories from fat. The Lean & Green meal is consumer selected and consists of 5-7 ounces of a lean protein, 1 ½ - 3 cups of non-starchy vegetables, and up to 2 healthy fat servings. The healthy snack(s) included in this plans consists of a consumer selected serving of grain/starch, dairy, or fruit.
  Groups: 5 & 2 & 2 Plan
Other: 4 & 2 & 1 Plan — Medifast has developed the 4 & 2 & 1 Plan as a higher calorie and higher carbohydrate alternative. This plan may be selected for very obese (BMI ≥ 40kg/m2) or older (>65 years) individuals, or for medical (e.g., diabetes) or behavioral reasons (individuals engages in high levels of physical activity). The 4 & 2 & 1 Plan consists of 4 Medifast meal replacements, 2 Lean & Green meals, and 1 healthy snack, providing 1,000-1,200 kcal, >72g protein, >100g carbohydrate, and <30% of calories from fat. The Lean & Green meal is consumer selected and consists of 5-7 ounces of a lean protein, 1 ½ - 3 cups of non-starchy vegetables, and up to 2 healthy fat servings. The healthy snack included in this plans consist of a consumer selected serving of grain/starch, dairy, or fruit.
  Groups: 4 & 2 & 1 Plan

SUMMARY:
The purpose of this study is to retrospectively and systematically review records of overweight and obese Medifast Weight Control Center (MWCC) members who have been assigned to the 5 & 2 & 2 Plan or the 4 & 2 & 1 Plan for weight loss to gain a better understanding of the effectiveness of these programs. The study will describe demographics of this population, along with weight loss, anthropometrics, body composition and effects on available cardiovascular parameters. Adherence to the plans will also be examined.

The study hypothesis is that the 5 & 2 & 2 Meal Replacement Plan and the 4 & 2 & 1 Meal Replacement Plan are both effective programs for weight loss in overweight and obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females, 18 years of age or older at the start of the weight loss program.
* Subject has a BMI ≥ 25 kg/m2.
* Subject started a weight management program at the MWCC location on or after January 1, 2012.
* Subject followed the 5 & 2 & 2 Plan or the 4 & 2 & 1 Plan for at least the first two weeks of their weight loss phase while an active member of the MWCC.
* Subject signed the Personal Health Information Consent Form.

Exclusion Criteria:

* Subject was concurrently following another weight loss program other than the 5 & 2 & 2 Plan or the 4 & 2 & 1 Plan while on that respective plan.
* Subject had documented use of prescription or over-the-counter weight loss pharmacotherapy (e.g., phentermine, Orlistat) concurrently with the 5 & 2 & 2 Plan or the 4 & 2 & 1 Plan.
* Subject completed initial consultation but did not participate in any follow-up visits.
* Subject is currently in the active weight loss phase of their program at the MWCC (Subjects in the transition or weight maintenance phases of their programs are eligible.)
* Written request by subject to revoke consent to use health information is present in subject chart.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is a systematic retrospective chart review of existing MWCC charts located in Maryland, Texas, Florida or Pennsylvania for MWCC members who used either the Medifast 5 & 2 & 2 Plan or the Medifast 4 & 2 & 1 Plan for weight loss.
  Charts will be reviewed for members that started either the 5 & 2 & 2 Plan or the 4 & 2 & 1 Plan on or after January 1, 2012. This start date was chosen because it represents the date when Medifast began using the current versions of the 5 & 2 & 2 Plan and the 4 & 2 & 1 Plan. Only charts of those members who are no longer in the active weight loss phase of their program at the MWCC will be considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda M Aterburn, PhD, Principal Investigator — Medifast, Inc.
Locations (1):
- Medifast, Inc., Owings Mills, Maryland, United States

REFERENCES:
- [Derived] Coleman CD, Kiel JR, Mitola AH, Langford JS, Davis KN, Arterburn LM. Effectiveness of a Medifast meal replacement program on weight, body composition and cardiometabolic risk factors in overweight and obese adults: a multicenter systematic retrospective chart review study. Nutr J. 2015 Aug 6;14:77. doi: 10.1186/s12937-015-0062-8. PMID 26245279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a retrospective chart review of Medifast Weight Control Center (MWCC) clients from 21 centers that used either the Medifast 5 & 2 & 2 Plan or 4 & 2 & 1 Plan for weight loss between 1/2012 and 3/2014 - it is retropsective and observational in nature, so there was no recruitment involved. The plans were evaluated separately and not compared.
Period: Overall Study
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Started | 62 (87 Charts were screened with 25 screen failures due to exclusion criteria.) | 310 (478 charts were screened with 168 screen failures due to exclusion criteria.)
Completed | 37 (There was no predefined study period to complete. 37 remained through the 12 wk primary endpoint.) | 185 (There was no predefined study period to complete. 185 remained through the 12 wk primary endpoint.)
Not Completed | 25 | 125

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan | Total
Number analyzed (Participants) | 62 | 310 | 372
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 222 | 277
  >=65 years | 7 | 88 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (13.7) | 53.5 (14.7) | 52.4 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 177 | 204
  Male | 35 | 133 | 168
Region of Enrollment [Number; unit: participants]
  United States | 62 | 310 | 372
Weight [Mean (Standard Deviation); unit: Pounds] | 327.11 (64.33) | 240.00 (47.83) | 254.02 (60.25)
BMI [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index
  kg/m2 | 48.7 (9.9) | 37.7 (6.8) | 39.5 (8.5)
Lean Body Mass [Mean (Standard Deviation); unit: Pounds] — Measured by bioelectrical impedance analysis
  Pounds | 168.52 (31.46) | 135.96 (31.24) | 140.33 (33.09)
Body Fat Mass [Mean (Standard Deviation); unit: Pounds] — Measured by bioelectrical impedance analysis
  Pounds | 152.46 (41.36) | 103.40 (30.58) | 110.04 (36.41)

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: The primary endpoint in this study is weight and the primary outcome is change from baseline body weight at 12 weeks for each plan (5 & 2 & 2 and 4 & 2 & 1 Plans). Change from baseline will also be examined at other predetermined time points (e.g., 1, 2, 4, 8, 16, 20 and 24 weeks, and final weight loss visit - the mean length of time from baseline to the final weight loss visit was 18.06 weeks for the 5 & 2 & 2 Plan and 17.35 weeks for the 4 & 2 & 1 Plan.).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 37 | 185
Pounds | -28.35 (15.60) | -23.95 (12.28)
Statistical Analysis 1: Comparison: 5 & 2 & 2 Plan vs 4 & 2 & 1 Plan; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Within group comparison (for each group) using a non-parametric paired Wilcoxon signed rank test comparing repeated measures in a single sample

2. Secondary Outcome: Percentage of Subjects Who Lose at Least 5% of Baseline Body Weight
Description: The categorical endpoint of the proportion of subjects who lose at least 5% of baseline body weight while on each plan (5 & 2 & 2 and 4 & 2 & 1 Plans).
Time Frame: 12 weeks
Measure: Number; unit: percentage of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 37 | 185
percentage of subjects | 75.7 | 85.4

3. Secondary Outcome: Proportion of Subjects Who Lose at Least 10% of Baseline Body Weight
Description: The categorical endpoint of the proportion of subjects who lose at least 10% of baseline body weight while on each program (5 & 2 & 2 and 4 & 2 & 1 Plans).
Time Frame: 12 weeks
Measure: Number; unit: percentage of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 37 | 185
percentage of subjects | 40.5 | 50.8

4. Secondary Outcome: Lean Mass
Description: Lean mass expressed as an absolute change from baseline.
Time Frame: 12 weeks
Population: Not all subjects remaining at 12 weeks had body composition testing performed.
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 12 | 86
Pounds | -5.47 (6.41) | -5.31 (4.89)

5. Secondary Outcome: Fat Mass
Description: Fat mass expressed as an absolute change from baseline.
Time Frame: 12 weeks
Population: Not all subjects remaining at 12 weeks had body composition testing performed.
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 12 | 86
Pounds | -21.09 (8.09) | -21.25 (10.90)

6. Secondary Outcome: Abdominal Circumference
Description: Abdominal circumference expressed as an absolute change from baseline.
Time Frame: 12 weeks
Population: Not all subjects remaining at 12 weeks had measurement performed.
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 10 | 73
Inches | -3.70 (1.30) | -4.47 (2.59)

7. Secondary Outcome: Waist Circumference
Description: Waist circumference expressed as an absolute change from baseline.
Time Frame: 12 weeks
Population: Not all subjects remaining at 12 weeks had measurement performed.
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 10 | 73
Inches | -3.55 (1.83) | -3.87 (2.34)

8. Secondary Outcome: Hip Circumference
Description: Hip circumference expressed as an absolute change from baseline.
Time Frame: 12 weeks
Population: Not all subjects remaining at 12 weeks had measurement performed.
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 10 | 73
Inches | -4.18 (2.96) | -3.41 (2.22)

9. Secondary Outcome: Blood Pressure
Description: Blood pressure (systolic and diastolic) expressed as an absolute change from baseline.
Time Frame: 12 weeks
Population: Not all subjects were remaining at 12 weeks and not all had measurement performed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 13 | 114
mmHg
  Systolic | -17.69 (17.61) | -11.27 (16.65)
  Diastolic | -8.38 (8.01) | -6.60 (12.62)

10. Secondary Outcome: Pulse
Description: Pulse expressed as an absolute change from baseline.
Time Frame: 12 weeks
Population: Not all subjects were remaining at 12 weeks and not all had measurement performed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 13 | 111
Beats per minute | -3.62 (10.04) | -2.95 (10.48)

11. Secondary Outcome: Blood Pressure Categorical
Description: Blood pressure expressed as a categorical variable (normotensive, pre-hypertensive and hypertensive based on National Institute of Health Guidelines) with the percent of participants that improved (e.g. from hypertensive to pre-hypertensive or normal) their blood pressure category from baseline to 12 weeks.
Time Frame: 12 weeks
Population: Not all subjects were remaining at 12 weeks and not all had measurement performed.
Measure: Number; unit: Percent of participants
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 13 | 114
Percent of participants | 53.8 | 49.1

12. Secondary Outcome: Resting Metabolic Rate
Description: Resting metabolic rate expressed as an absolute change from baseline to final weight loss visit (The average length of time from baseline to the final weight loss visit was 18 weeks for the 5 & 2 & 2 Plan and 17 weeks for the 4 & 2 & 1 Plan.).
Time Frame: Baseline to final weight loss visit (Average of 18 weeks for the 5 & 2 & 2 Plan and 17 weeks for the 4 & 2 & 1 Plan)
Population: Number of participants with paired data at baseline and final weight loss visit was too small for meaningful analysis.
Measure: Mean (Standard Deviation); unit: calories
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 1 | 6
calories | 10 (0) | -216.67 (279.48)

13. Secondary Outcome: Adherence
Description: Adherence will be assessed through attendance at weekly visits and documented use of meal replacements at each visit. (Meal replacement adherence=average number of self-reported daily meal replacements through 12 weeks/nuber of prescribed meal replacements; Attendance adherence=number of visits/number of weeks on plan
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percent Compliant
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 62 | 310
Percent Compliant
  Meal replacement compliance | 83.85 (16.67) | 88.79 (18.64)
  Attendance compliance | 83.65 (19.09) | 85.71 (17.94)

14. Secondary Outcome: Proportion of Subjects Who Lose at Least 5% of Baseline Body Weight
Description: as for outcome 2
Time Frame: 1 weeks
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 54 | 283
Percent of subjects | 1.6 | 3.2

15. Secondary Outcome: Proportion of Subjects Who Lose at Least 5% of Baseline Body Weight
Description: as for outcome 2
Time Frame: 2 weeks
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 56 | 280
Percent of subjects | 8.9 | 16.1

16. Secondary Outcome: Proportion of Subjects Who Lose at Least 5% of Baseline Body Weight
Description: as for outcome 2
Time Frame: 4 weeks
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 57 | 289
Percent of subjects | 33.3 | 50.2

17. Secondary Outcome: Proportion of Subjects Who Lose at Least 5% of Baseline Body Weight
Description: as for outcome 2
Time Frame: 8 weeks
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 48 | 239
Percent of subjects | 72.9 | 76.2

18. Secondary Outcome: Proportion of Subjects Who Lose at Least 5% of Baseline Body Weight
Description: as for outcome 2
Time Frame: 16 weeks
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 24 | 151
Percent of subjects | 95.8 | 92.7

19. Secondary Outcome: Proportion of Subjects Who Lose at Least 5% of Baseline Body Weight
Description: as for outcome 2
Time Frame: 20 weeks
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 23 | 112
Percent of subjects | 95.7 | 94.6

20. Secondary Outcome: Proportion of Subjects Who Lose at Least 5% of Baseline Body Weight
Description: as for outcome 2
Time Frame: 24 weeks
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 17 | 81
Percent of subjects | 88.2 | 96.3

21. Secondary Outcome: Proportion of Subjects Who Lose at Least 5% of Baseline Body Weight
Description: The categorical endpoint of the proportion of subjects who lose at least 5% of baseline body weight while on each plan (5 & 2 & 2 and 4 & 2 & 1 Plans) at their final weight loss visit (The mean length of time from baseline to the final weight loss visit was 18 weeks for the 5 & 2 & 2 Plan and 17 weeks for the 4 & 2 & 1 Plan.).
Time Frame: Baseline to final weight loss visit (Average of 18 weeks for the 5 & 2 & 2 Plan and 17 weeks for the 4 & 2 & 1 Plan)
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 62 | 306
Percent of subjects | 62.9 | 69.6

22. Secondary Outcome: Proportion of Subjects Who Lose at Least 10% of Baseline Body Weight
Description: as for outcome 3
Time Frame: 1 weeks
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 54 | 283
Percent of subjects | 0.0 | 0.0

23. Secondary Outcome: Proportion of Subjects Who Lose at Least 10% of Baseline Body Weight
Description: as for outcome 3
Time Frame: 2 weeks
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 56 | 280
Percent of subjects | 0.0 | 0.0

24. Secondary Outcome: Proportion of Subjects Who Lose at Least 10% of Baseline Body Weight
Description: as for outcome 3
Time Frame: 4 weeks
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 57 | 289
Percent of subjects | 0.0 | 1.0

25. Secondary Outcome: Proportion of Subjects Who Lose at Least 10% of Baseline Body Weight
Description: as for outcome 3
Time Frame: 8 weeks
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 48 | 239
Percent of subjects | 16.7 | 23.0

26. Secondary Outcome: Proportion of Subjects Who Lose at Least 10% of Baseline Body Weight
Description: as for outcome 3
Time Frame: 16 weeks
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 24 | 151
Percent of subjects | 50.0 | 64.9

27. Secondary Outcome: Proportion of Subjects Who Lose at Least 10% of Baseline Body Weight
Description: as for outcome 3
Time Frame: 20 weeks
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 23 | 112
Percent of subjects | 56.5 | 69.6

28. Secondary Outcome: Proportion of Subjects Who Lose at Least 10% of Baseline Body Weight
Description: as for outcome 3
Time Frame: 24 weeks
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 17 | 81
Percent of subjects | 58.8 | 75.3

29. Secondary Outcome: Proportion of Subjects Who Lose at Least 10% of Baseline Body Weight
Description: The categorical endpoint of the proportion of subjects who lose at least 10% of baseline body weight while on each program (5 & 2 & 2 and 4 & 2 & 1 Plans) at their final weight loss visit (The mean length of time from baseline to the final weight loss visit was 18 weeks for the 5 & 2 & 2 Plan and 17 weeks for the 4 & 2 & 1 Plan.).
Time Frame: Baseline to final weight loss visit (Average of 18 weeks for the 5 & 2 & 2 Plan and 17 weeks for the 4 & 2 & 1 Plan)
Measure: Number; unit: Percent of subjects
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 62 | 306
Percent of subjects | 29.0 | 39.9

30. Secondary Outcome: Lean Mass
Description: Lean mass expressed as an absolute change from baseline.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 26 | 177
Pounds | -5.19 (5.42) | -4.50 (4.66)

31. Secondary Outcome: Lean Mass
Description: Lean mass expressed as an absolute change from baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 11 | 96
Pounds | -8.36 (5.67) | -4.49 (5.36)

32. Secondary Outcome: Lean Mass
Description: Lean mass expressed as an absolute change from baseline.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 8 | 55
Pounds | -11.15 (4.62) | -4.29 (6.45)

33. Secondary Outcome: Lean Mass
Description: Lean mass expressed as an absolute change from baseline.
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 6 | 44
Pounds | -13.83 (5.33) | -5.08 (6.96)

34. Secondary Outcome: Lean Mass
Description: Lean mass expressed as an absolute change from baseline.
Time Frame: 24 weeks
Population: Not all subjects were remaining at 24 weeks and not all had measurement performed.
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 3 | 55
Pounds | -14.35 (9.14) | -6.79 (6.45)

35. Secondary Outcome: Fat Mass
Description: Fat mass expressed as an absolute change from baseline.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 26 | 177
Pounds | -11.46 (6.92) | -9.09 (7.71)

36. Secondary Outcome: Fat Mass
Description: Fat mass expressed as an absolute change from baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 11 | 106
Pounds | -17.35 (5.80) | -16.27 (8.16)

37. Secondary Outcome: Fat Mass
Description: Fat mass expressed as an absolute change from baseline.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 8 | 70
Pounds | -26.38 (9.11) | -26.34 (12.16)

38. Secondary Outcome: Fat Mass
Description: Fat mass expressed as an absolute change from baseline.
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 6 | 53
Pounds | -34.03 (11.64) | -29.03 (17.00)

39. Secondary Outcome: Abdominal Circumference
Description: Abdominal circumference expressed as an absolute change from baseline.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 27 | 158
Inches | -2.81 (2.08) | -1.86 (1.71)

40. Secondary Outcome: Abdominal Circumference
Description: Abdominal circumference expressed as an absolute change from baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 16 | 86
Inches | -4.42 (3.04) | -3.28 (1.99)

41. Secondary Outcome: Abdominal Circumference
Description: Abdominal circumference expressed as an absolute change from baseline.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 6 | 63
Inches | -5.71 (1.19) | -4.46 (2.73)

42. Secondary Outcome: Abdominal Circumference
Description: Abdominal circumference expressed as an absolute change from baseline.
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 7 | 41
Inches | -6.25 (1.89) | -5.78 (3.06)

43. Secondary Outcome: Abdominal Circumference
Description: Abdominal circumference expressed as an absolute change from baseline.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 3 | 24
Inches | -4.83 (5.16) | -5.98 (2.74)

44. Secondary Outcome: Waist Circumference
Description: Waist circumference expressed as an absolute from baseline.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 27 | 158
Inches | -2.21 (1.49) | -1.97 (1.37)

45. Secondary Outcome: Waist Circumference
Description: Waist circumference expressed as an absolute change from baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 16 | 86
Inches | -3.60 (2.42) | -3.24 (1.72)

46. Secondary Outcome: Waist Circumference
Description: Waist circumference expressed as an absolute change from baseline.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 6 | 63
Inches | -4.38 (2.06) | -4.75 (2.22)

47. Secondary Outcome: Waist Circumference
Description: Waist circumference expressed as an absolute change from baseline.
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 7 | 41
Inches | -6.93 (2.49) | -5.32 (2.70)

48. Secondary Outcome: Waist Circumference
Description: Waist circumference expressed as an absolute change from baseline.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 3 | 24
Inches | -3.92 (3.89) | -5.35 (2.88)

49. Secondary Outcome: Hip Circumference
Description: Hip circumference expressed as an absolute change from baseline.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 27 | 158
Inches | -2.40 (1.88) | -1.56 (1.36)

50. Secondary Outcome: Hip Circumference
Description: Hip circumference expressed as an absolute change from baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 14 | 86
Inches | -3.34 (1.99) | -2.68 (1.64)

51. Secondary Outcome: Hip Circumference
Description: Hip circumference expressed as an absolute change from baseline.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 6 | 63
Inches | -4.42 (3.02) | -3.97 (2.15)

52. Secondary Outcome: Hip Circumference
Description: Hip circumference expressed as an absolute change from baseline.
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 6 | 41
Inches | -5.38 (1.90) | -5.38 (3.96)

53. Secondary Outcome: Hip Circumference
Description: Hip circumference expressed as an absolute change from baseline.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 3 | 24
Inches | -5.17 (3.33) | -4.92 (2.68)

54. Secondary Outcome: Blood Pressure
Description: Blood pressure (systolic and diastolic) expressed as an absolute change from baseline.
Time Frame: 1 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 24 | 165
mmHg
  Systolic | -4.63 (17.17) | -5.80 (14.05)
  Diastolic | -2.63 (10.49) | -3.59 (9.98)

55. Secondary Outcome: Blood Pressure
Description: Blood pressure (systolic and diastolic) expressed as an absolute change from baseline.
Time Frame: 2 weeks
Population: Not all subjects were remaining at 2 weeks and not all had measurement performed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 22 | 174
mmHg
  Systolic | -6.41 (15.63) | -8.53 (13.97)
  Diastolic | -2.91 (9.89) | -5.37 (10.84)

56. Secondary Outcome: Blood Pressure
Description: Blood pressure (systolic and diastolic) expressed as an absolute change from baseline.
Time Frame: 4 weeks
Population: Not all subjects were remaining at 4 weeks and not all had measurement performed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 26 | 175
mmHg
  Systolic | -7.81 (19.76) | -9.87 (16.93)
  Diastolic | -7.31 (9.00) | -5.90 (12.13)

57. Secondary Outcome: Blood Pressure
Description: Blood pressure (systolic and diastolic) expressed as an absolute change from baseline.
Time Frame: 8 weeks
Population: Not all subjects were remaining at 8 weeks and not all had measurement performed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 24 | 144
mmHg
  Systolic | -14.21 (26.06) | -7.51 (14.68)
  Diastolic | -9.25 (11.30) | -6.11 (11.09)

58. Secondary Outcome: Blood Pressure
Description: Blood pressure (systolic and diastolic) expressed as an absolute change from baseline.
Time Frame: 16 weeks
Population: Not all subjects were remaining at 16 weeks and not all had measurement performed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 11 | 95
mmHg
  Systolic | -19.27 (25.09) | -10.59 (17.03)
  Diastolic | -8.55 (11.60) | -6.84 (9.94)

59. Secondary Outcome: Blood Pressure
Description: Blood pressure (systolic and diastolic) expressed as an absolute change from baseline.
Time Frame: 20 weeks
Population: Not all subjects were remaining at 20 weeks and not all had measurement performed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 11 | 70
mmHg
  Systolic | -21.55 (20.62) | -9.34 (17.49)
  Diastolic | -8.55 (11.12) | -6.26 (13.05)

60. Secondary Outcome: Blood Pressure
Description: Blood pressure (systolic and diastolic) expressed as an absolute change from baseline.
Time Frame: 24 weeks
Population: Not all subjects were remaining at 24 weeks and not all had measurement performed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 9 | 52
mmHg
  Systolic | -14.33 (16.19) | -7.79 (19.40)
  Diastolic | -5.44 (8.41) | -3.92 (14.18)

61. Secondary Outcome: Blood Pressure
Description: Blood pressure (systolic and diastolic) expressed as an absolute change from baseline to final weight loss visit (The mean length of time from baseline to the final weight loss visit was 18 weeks for the 5 & 2 & 2 Plan and 17 weeks for the 4 & 2 & 1 Plan.).
Time Frame: Baseline to final weight loss visit (Average of 18 weeks for the 5 & 2 & 2 Plan and 17 weeks for the 4 & 2 & 1 Plan)
Population: Not all subjects had measurement performed at their final visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 24 | 163
mmHg
  Systolic | -16.96 (21.79) | -9.52 (15.62)
  Diastolic | -7.08 (10.68) | -5.64 (11.58)

62. Secondary Outcome: Pulse
Description: Pulse expressed as an absolute change from baseline.
Time Frame: 1 weeks
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 24 | 162
Beats per minute | -0.46 (12.86) | 1.07 (9.42)

63. Secondary Outcome: Pulse
Description: Pulse expressed as an absolute change from baseline.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 22 | 173
mmHg | -3.27 (10.27) | -1.21 (9.94)

64. Secondary Outcome: Pulse
Description: Blood pressure (systolic and diastolic) expressed as an absolute change from baseline.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 26 | 175
Beats per minute | -1.62 (12.52) | -2.88 (10.11)

65. Secondary Outcome: Pulse
Description: Pulse expressed as an absolute change from baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 24 | 142
Beats per minute | -1.17 (17.84) | -2.65 (10.71)

66. Secondary Outcome: Pulse
Description: Pulse expressed as an absolute change from baseline.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 11 | 95
Beats per minute | -3.27 (11.29) | -3.73 (11.89)

67. Secondary Outcome: Pulse
Description: Pulse expressed as an absolute change from baseline.
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 11 | 71
Beats per minute | 0.27 (13.27) | -2.31 (11.78)

68. Secondary Outcome: Pulse
Description: Pulse expressed as an absolute change from baseline.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 9 | 51
Beats per minute | 0.00 (4.66) | -3.67 (9.34)

69. Secondary Outcome: Pulse
Description: Pulse expressed as an absolute change from baseline to final weight loss visit (The mean length of time from baseline to the final weight loss visit was 18 weeks for the 5 & 2 & 2 Plan and 17 weeks for the 4 & 2 & 1 Plan.).
Time Frame: Baseline to final weight loss visit (Average of 18 weeks for the 5 & 2 & 2 Plan and 17 weeks for the 4 & 2 & 1 Plan)
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 24 | 161
Beats per minute | -2.29 (10.75) | -2.29 (11.63)

70. Secondary Outcome: Adherence
Description: Adherence will be assessed through documented use of meal replacements at each visit.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Percent compliance meal replacements
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 53 | 276
Percent compliance meal replacements | 94.53 (13.09) | 96.29 (14.45)

71. Secondary Outcome: Adherence
Description: Adherence will be assessed through documented use of meal replacements at each visit.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Percent compliance meal replacements
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 47 | 225
Percent compliance meal replacements | 88.3 (20.99) | 95.17 (14.97)

72. Secondary Outcome: Adherence
Description: Adherence will be assessed through documented use of meal replacements at each visit.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Percent compliance meal replacements
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 21 | 145
Percent compliance meal replacements | 79.52 (26.55) | 94.29 (17.19)

73. Secondary Outcome: Adherence
Description: Adherence will be assessed through documented use of meal replacements at each visit.
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: Percent compliance meal replacements
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 20 | 107
Percent compliance meal replacements | 89.00 (18.04) | 89.25 (26.79)

74. Secondary Outcome: Adherence
Description: Adherence will be assessed through documented use of meal replacements at each visit.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Percent compliance meal replacements
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 15 | 74
Percent compliance meal replacements | 90.67 (14.86) | 91.22 (23.47)

75. Secondary Outcome: Adherence
Description: Adherence will be assessed through documented use of meal replacements at each visit from baseline (The mean length of time from baseline to the final weight loss visit was 18 weeks for the 5 & 2 & 2 Plan and 17 weeks for the 4 & 2 & 1 Plan.).
Time Frame: Baseline to final weight loss visit (Average of 18 weeks for the 5 & 2 & 2 Plan and 17 weeks for the 4 & 2 & 1 Plan)
Measure: Mean (Standard Deviation); unit: Percent compliance meal replacements
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 58 | 273
Percent compliance meal replacements | 82.41 (27.49) | 85.26 (29.43)

76. Secondary Outcome: Body Weight
Description: Change in body weight from baseline reported as absolute change.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 54 | 283
Pounds | -7.64 (4.86) | -5.95 (3.33)

77. Secondary Outcome: Body Weight
Description: Change in body weight from baseline reported as absolute change from baseline.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 56 | 280
Pounds | -9.71 (4.95) | -8.24 (4.27)

78. Secondary Outcome: Body Weight
Description: Change in body weight from baseline reported absolute change from baseline.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 57 | 289
Pounds | -14.26 (6.88) | -12.25 (6.01)

79. Secondary Outcome: Body Weight
Description: Change in body weight from baseline reported as absolute change.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Pound
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 48 | 239
Pound | -22.81 (11.21) | -18.32 (9.21)

80. Secondary Outcome: Body Weight
Description: Change in body weight from baseline reported as absolute change.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 24 | 151
Pounds | -36.89 (16.45) | -28.84 (14.48)

81. Secondary Outcome: Body Weight
Description: Change in body weight from baseline reported as absolute change.
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 23 | 112
Pounds | -40.51 (19.08) | -32.42 (16.22)

82. Secondary Outcome: Body Weight
Description: Change in body weight from baseline to final weight loss visit reported as absolute change. (The mean length of time from baseline to the final weight loss visit was 18 weeks for the 5 & 2 & 2 Plan and 17 weeks for the 4 & 2 & 1 Plan.)
Time Frame: Baseline to final weight loss visit (Average of 18 weeks for the 5 & 2 & 2 Plan and 17 weeks for the 4 & 2 & 1 Plan)
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 62 | 306
Pounds | -29.25 (27.65) | -23.34 (18.65)

83. Secondary Outcome: Fat Mass
Description: Fat mass expressed as an absolute change from baseline.
Time Frame: 24 weeks
Population: Not all subjects remaining at 24 weeks had body composition testing performed.
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
Number analyzed (Participants) | 4 | 35
Pounds | -56.88 (18.52) | -32.00 (15.76)

ADVERSE EVENTS:
Time Frame: Charts from MWCC customers that followed either the 5 & 2 & 2 Plan or the 4 & 2 & 1 Plan and met inclusion criteria who started their weight loss plan on or after January 1, 2012 and completed the active weight loss phase of their plan by March 31, 2014 (a total period of 2 years and 3 months).
Description: This is a retrospective chart review study, and all of the signs, symptoms, and incidents reported were lay accounts by MWCC staff during the routine visits that were included as a part of customers' weight loss programs - not specifically as part of a clinical trial. Therefore, information normally associated with adverse events (relatedness, seriousness, etc.) was not collected. This description pertains to all events (all-cause mortality, serious adverse events, and other adverse events.
Arm/Group | 5 & 2 & 2 Plan | 4 & 2 & 1 Plan
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/310
Serious Adverse Events (participants affected / at risk) | 2/62 | 9/310
Other Adverse Events (participants affected / at risk) | 46/62 | 219/310
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 & 2 & 2 Plan (N=62) | 4 & 2 & 1 Plan (N=310)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
Heart attack (Cardiac disorders) | 0 (0) | 1 (1)
cholecystectomy (Surgical and medical procedures) | 1 (1) | 2 (2)
Bloot clot (Vascular disorders) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 0 (0) | 1 (1)
Ruptured hemorrhoid (Surgical and medical procedures) | 0 (0) | 1 (1)
Mini-stroke (Vascular disorders) | 1 (1) | 0 (0)
Hospitalization (General disorders) | 0 (0) | 2 (2) — Reason for hospitalizations was not specified in these 2 cases.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 & 2 & 2 Plan (N=62) | 4 & 2 & 1 Plan (N=310)
constipation (Gastrointestinal disorders) | 9 (9) | 33 (33)
gas/bloating (Gastrointestinal disorders) | 1 (1) | 22 (22)
hunger (General disorders) | 12 (12) | 56 (56)
fatigue (General disorders) | 3 (3) | 34 (34)
stress/anxiety (General disorders) | 5 (5) | 16 (16)
Sick Not Otherwise Specified (General disorders) | 13 (13) | 69 (69)
cravings (General disorders) | 5 (5) | 14 (14)
Headache (General disorders) | 6 (6) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes